CLINICAL TRIAL: NCT07273591
Title: Effects of Low-level Laser Therapy on Spasticity and Gait Parameters in Chronic Stroke Patients With Spastic Plantar Flexors
Acronym: LLLT-STROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montiha Azeem (Other)
Responsible Party: Sponsor-Investigator, Montiha Azeem, Principal Investigator, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-UOL-/544-08/24
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Spasticity; Plantar Flexors
Keywords: Chronic stroke; Low-level LASER therapy; planter flexors; spasticity; gait abnormalities
MeSH Terms: conditions — Stroke; Muscle Spasticity; Mobility Limitation | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy (Active Comparator): Participants in control group received conventional physical therapy for spasticity that was consisted of heating modality for 20 minutes followed by ten repetitions of sustained stretching of calf muscles (10 seconds hold), strengthening exercise for lower limb muscles i.e. calf muscles, hamstrings, and quadriceps, balance training on balance board and training of gait in parallel bars and using the stepper for six weeks and three sessions each week
  Interventions: Other: conventional physical therapy
- low level laser therapy (Experimental): Patients were in prone position while we applied low level laser therapy in continues wave at a wavelength in the near infrared of 830nm. Power density was 670 mW/cm2. The treatment time per point was 30 seconds. Probe head was placed at 90 degree with light pressure on the calf muscles. Three consecutive treatments were given in a session, with 5 seconds break in between, giving a total irradiation time of 90 seconds. Three sessions were given per week for total of six weeks
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Low Level Laser Therapy — Patients were in prone position while we applied low level laser therapy in continues wave at a wavelength in the near infrared of 830nm. Power density was 670 mW/cm2. The treatment time per point was 30 seconds. Probe head was placed at 90 degree with light pressure on the calf muscles. Three consecutive treatments were given in a session, with 5 seconds break in between, giving a total irradiation time of 90 seconds. Three sessions were given per week for total of six weeks
  Other Names: LLLT; Infrared laser therapy; photobiomodulation
  Arms: low level laser therapy
Other: conventional physical therapy — Participants in control group received conventional physical therapy for spasticity that was consisted of heating modality for 20 minutes followed by ten repetitions of sustained stretching of calf muscles (10 seconds hold), strengthening exercise for lower limb muscles i.e. calf muscles, hamstrings, and quadriceps, balance training on balance board and training of gait in parallel bars and using the stepper for six weeks and three sessions each week.
  Other Names: routine physiotherapy; traditional physical therapy
  Arms: conventional physical therapy

SUMMARY:
Stroke is one of the leading causes of long-term disability worldwide. Many patients who survive a stroke experience muscle stiffness (called spasticity), especially in the ankle and foot muscles, which makes walking difficult and painful. Spasticity in the plantar flexor muscles those that help push the foot down can lead to poor balance, limited mobility, and increased risk of falls.

This study aims to explore the effects of low-level laser therapy (LLLT) on spasticity and walking ability in patients who have had a stroke for more than six months (chronic stroke). LLLT is a non-invasive, painless treatment that uses low-intensity light to stimulate tissue healing, reduce muscle tightness, and improve nerve function.

A total of 18 chronic stroke patients with spastic plantar flexors were included in this randomized controlled trial (RCT). Participants were randomly assigned to one of two groups:

Study group: Received low-level laser therapy along with conventional physiotherapy.

Control group: Received conventional physiotherapy alone. Each patient received therapy for three weeks. The study evaluated outcomes using the Modified Ashworth Scale (MAS) for muscle spasticity, the Wisconsin Gait Scale (WGS) for walking quality, and a Goniometer for ankle joint range of motion. Assessments were done before and after treatment.

The results showed that both groups improved significantly, but patients who received laser therapy demonstrated greater reduction in spasticity and better gait performance compared to those who received conventional therapy alone.

This study suggests that low-level laser therapy can be a useful addition to conventional rehabilitation programs for improving walking ability and reducing spasticity in stroke patients.

DETAILED DESCRIPTION:
Background and Rationale:

After a stroke, damage to the brain can cause increased muscle tone (spasticity), reduced mobility, and altered gait patterns. These issues significantly affect independence and quality of life. Traditional physiotherapy techniques, such as stretching and strengthening, are helpful but often insufficient in chronic cases. Recent evidence suggests that low-level laser therapy (LLLT) can promote cellular recovery, improve blood circulation, and reduce muscle stiffness by enhancing nerve conduction and reducing inflammation.

Study Objective:

To determine the effectiveness of low-level laser therapy in improving spasticity and gait parameters in chronic stroke patients with spastic plantar flexors.

Study Design:

This was a randomized controlled trial conducted on 18 participants diagnosed with chronic stroke and presenting with spasticity of the ankle plantar flexors. Participants were divided into:

Study group (n=9): Received low-level laser therapy (parameters: wavelength 830 nm, power output 50 mW, energy density 6 J/cm²) combined with conventional physiotherapy.

Control group (n=9): Received conventional physiotherapy only (stretching, strengthening, and gait training).

Intervention Duration:

Both groups received treatment sessions five times a week for three weeks.

Outcome Measures:

Spasticity: Measured using the Modified Ashworth Scale (MAS) Gait Parameters: Measured using the Wisconsin Gait Scale (WGS) Ankle Range of Motion (ROM): Measured with a Goniometer

Data Analysis:

Within-group changes were assessed using Friedman's test, and between-group comparisons were made using the Mann-Whitney U test. A p-value ≤ 0.05 was considered statistically significant. Statistical analysis was performed using SPSS version 25.

Results Summary:

Both groups showed significant improvements in spasticity, ankle range of motion, and gait scores; however, the study group demonstrated greater gains in all parameters. The combination of LLLT with physiotherapy enhanced motor control, reduced stiffness, and improved walking quality more effectively than physiotherapy alone.

Conclusion:

Low-level laser therapy is a safe, effective, and non-invasive intervention that significantly improves spasticity and gait in chronic stroke patients. Incorporating LLLT into rehabilitation programs may help enhance mobility and functional independence.

ELIGIBILITY:
Inclusion Criteria:

Patients with Age of 45-70 years. Male and female patients with chronic stroke. Patients determined to have persistent stroke for no less than 1 year A maximum of 2 degrees of plantar flexor spasticity on MAS. (35) Cognitive preserved, having score of 24 to 30 on MMSE. (25) Medical referral for physiotherapy.

Exclusion Criteria:

Patients with uncontrolled metabolic illnesses, orthopedic issues, and other neurologic abnormalities should be excluded as potential confounding factors impacting balance performance. Patients with recurrent stroke. Patients who were at that point performing organized proactive tasks, for example, muscle reinforcing works out, Pilates, yoga or focused energy oxygen consuming activities Patients with Hypoesthesia or possibly Hyperesthesia of the side to be analyzed.

The patients with active contamination and presence of rashes at the site of utilization of the laser application. A neoplastic lesion at the site of application.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Change in Spasticity of Ankle Plantar Flexors Measured by Modified Ashworth Scale (MAS) | 6 weeks
  Spasticity of the ankle plantar flexors will be assessed using the Modified Ashworth Scale (MAS), a standardized clinical measure of muscle tone. Scores range from 0 (no increase in tone) to 4 (rigid in flexion or extension). Measurements will be taken at baseline, at 3 weeks, and at 6 weeks after the start of intervention. A decrease in MAS score will indicate improvement in spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Montiha Azeem, DPT, Principal Investigator — The University of Lahore, Lahore
Locations (1):
- Shalamar Hospital, Sughra Shafi Medical Complex, Narowal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No